CLINICAL TRIAL: NCT04754321
Title: HNSALV Trial: Combining Immunotherapy With Salvage Surgery and IORT for Treatment of Persistent/Recurrent Head and Neck Cancers
Brief Title: Combining Immunotherapy Salvage Surgery & IORT Tx Persistent/Recurrent Head & Neck Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Dukagjin Blakaj, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20297; NCI-2021-00036 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Carcinoma of Unknown Primary; Locally Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Pharyngeal Squamous Cell Carcinoma; Resectable Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiation; Radiotherapy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (pembrolizumab, salvage surgery, IORT) (Experimental): Patients receive pembrolizumab IV on day 1 of week 1, and undergo salvage surgery during week 4. Beginning week 8, patients receive pembrolizumab IV every 3 weeks for up to 18 doses in the absence of disease progression or unacceptable toxicity. Patients also undergo IORT for 1 fraction during week 9. Treatment with pembrolizumab may continue beyond initial progression per investigator-assessed clinical benefit and if the patient is tolerating pembrolizumab.
  Interventions: Radiation: Intraoperative Radiation Therapy; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Procedure: Salvage Surgery
- Arm B (pembrolizumab, EBRT, salvage surgery, IORT) (Experimental): Patients receive pembrolizumab IV on day 1 of week 1, and undergo low dose EBRT for 2 fractions on 2 consecutive days during week 4. Patients also undergo salvage surgery during week 8. Beginning week 11, patients receive pembrolizumab IV every 3 weeks for up to 18 doses in the absence of disease progression or unacceptable toxicity. Patients also undergo IORT for 1 fraction during week 11. Treatment with pembrolizumab may continue beyond initial progression per investigator-assessed clinical benefit and if the patient is tolerating pembrolizumab.
  Interventions: Radiation: External Beam Radiation Therapy; Radiation: Intraoperative Radiation Therapy; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Procedure: Salvage Surgery
- Arm C (pembrolizumab, EBRT, salvage surgery, IORT) (Experimental): Patients receive pembrolizumab IV on day 1 of week 1, and undergo high dose EBRT for 2 fractions on 2 consecutive days during week 4. Patients also undergo salvage surgery during week 8. Beginning week 11, patients receive pembrolizumab IV every 3 weeks for up to 18 doses in the absence of disease progression or unacceptable toxicity. Patients also undergo IORT for 1 fraction during week 11. Treatment with pembrolizumab may continue beyond initial progression per investigator-assessed clinical benefit and if the patient is tolerating pembrolizumab.
  Interventions: Radiation: External Beam Radiation Therapy; Radiation: Intraoperative Radiation Therapy; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Procedure: Salvage Surgery

INTERVENTIONS:
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam
  Arms: Arm B (pembrolizumab, EBRT, salvage surgery, IORT); Arm C (pembrolizumab, EBRT, salvage surgery, IORT)
Radiation: Intraoperative Radiation Therapy — Undergo IORT
  Other Names: Intraoperative Radiotherapy; IORT; radiotherapy, intraoperative
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Salvage Surgery — Undergo salvage surgery
  Other Names: Rescue Surgery; Salvage Resection; Salvage Surgical Resection; Surgical Salvage

SUMMARY:
This phase I trial is to find out the possible side effects of pembrolizumab and radiation therapy before and during surgery in treating patients with head and neck squamous cell cancer that remains despite treatment (persistent) or has come back (recurrent). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays or protons to kill tumor cells and shrink tumors. Giving pembrolizumab and radiation therapy before and during surgery may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the potential toxicity of immunotherapy and preoperative radiation combined with intra-operative radiation in patients with recurrent or persistent head and neck squamous cell carcinoma (HNSCC).

SECONDARY OBJECTIVES:

I. To evaluate the clinical efficacy, measured as a locoregional control rate (LCR) and progression-free survival (PFS), of immunotherapy and preoperative radiation combined with intra-operative radiation in patients with recurrent or persistent HNSCC.

II. To evaluate the pre-operative radiation dose effect (0 Gy, 2 Gy X 2, 8 Gy X 2) on anti-tumor immune response in the setting of immunotherapy in patients with recurrent or persistent HNSCC.

III. To evaluate the radiation dose effect (0 Gy, 2 Gy X 2, 8 Gy X 2) on the expression of the deoxyribonucleic acid (DNA) exonuclease Trex1.

IV. To compare the overall survival (OS) of pembrolizumab and pre and post-operative external beam radiation therapy (EBRT) plus intraoperative radiation therapy (IORT) in subjects with recurrent or persistent HNSCC.

V. To assess the overall safety and tolerability of pre-operative pembrolizumab and pre-operative EBRT and IORT plus post-operative pembrolizumab versus pre-operative pembrolizumab plus IORT and post-operative pembrolizumab in subjects with with recurrent or persistent HNSCC.

VI. To evaluate whether PD-L1 expression is a predictive biomarker for LCR and PFS.

VII. To evaluate whether TNF-alpha expression is a predictive biomarker for LCR and PFS.

VIII. To evaluate whether NFkappaB expression is a predictive biomarker for LCR and PFS.

IX. To evaluate whether tumor mutational burden is predictive of immunotherapy response.

X. To evaluate the Health Related Quality of Life (HRQoL) as assessed by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core 30 (QLQ-C30) and QLQ-HN35.

EXPLORATORY OBJECTIVES:

I. To evaluate associations between gene expression status of tumor samples and clinical efficacy (LRC, PFS and overall survival [OS]).

II. To evaluate whether mutational burden is a predictive biomarker for LCR and PFS.

III. To explore potential biomarkers associated with clinical efficacy (LRC, PFS, and OS) by analyzing circulating tumor DNA quantitative load with polymerase chain reaction (PCR), chemokines/cytokines and immune cells (e.g. CD8+ T cells, regulatory T cells [Tregs], myeloid derived suppressor cells [MDSCs]) with FACS in blood, tumor tissue and correlating those with clinical outcomes.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM A: Patients receive pembrolizumab intravenously (IV) on day 1 of week 1, and undergo salvage surgery during week 4. Beginning week 8, patients receive pembrolizumab IV every 3 weeks for up to 18 doses in the absence of disease progression or unacceptable toxicity. Patients also undergo intraoperative radiation therapy (IORT) for 1 fraction during week 9. Treatment with pembrolizumab may continue beyond initial progression per investigator-assessed clinical benefit and if the patient is tolerating pembrolizumab.

ARM B: Patients receive pembrolizumab IV on day 1 of week 1, and undergo low dose EBRT for 2 fractions on 2 consecutive days during week 4. Patients also undergo salvage surgery during week 8. Beginning week 11, patients receive pembrolizumab IV every 3 weeks for up to 18 doses in the absence of disease progression or unacceptable toxicity. Patients also undergo IORT for 1 fraction during week 11. Treatment with pembrolizumab may continue beyond initial progression per investigator-assessed clinical benefit and if the patient is tolerating pembrolizumab.

ARM C: Patients receive pembrolizumab IV on day 1 of week 1, and undergo high dose EBRT for 2 fractions on 2 consecutive days during week 4. Patients also undergo salvage surgery during week 8. Beginning week 11, patients receive pembrolizumab IV every 3 weeks for up to 18 doses in the absence of disease progression or unacceptable toxicity. Patients also undergo IORT for 1 fraction during week 11. Treatment with pembrolizumab may continue beyond initial progression per investigator-assessed clinical benefit and if the patient is tolerating pembrolizumab.

After completion of study treatment, patients are followed up at 90 and 180 days, then every 90 weeks for 24 months, and then every 6 months up to year 5.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed either persistent and/ or locoregionally recurrent HNSCC of oral cavity, pharynx, larynx, unknown primary head and neck (H&N) squamous cell carcinoma
* Resectable disease as determined by the surgeon and team
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) < 2
* At least 18 years of age
* Adequate hematologic, renal, and hepatic function
* Must have at least 2 week washout period from prior therapy
* Willingness and ability to provide informed consent
* Negative pregnancy test for females of reproductive potential
* Patients who have undergone therapy for their cancer, such as surgery and/or chemotherapy and/or radiotherapy and recurred
* Disease measurable by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1 criteria.
* Prior definitive and palliative chemotherapy will be allowed
* Prior radiation therapy will be allowed
* Tumor tissue from resected site of disease must be provided for biomarker analyses, in addition to urine and blood sample as scheduled per protocol
* White blood cell (WBC) >= 2000/uL (obtained within 14 days of randomization)
* Neutrophils >= 1500/uL (obtained within 14 days of randomization)
* Platelets >= 100 x10^3/uL (obtained within 14 days of randomization)
* Hemoglobin > 9.0 g/dL (obtained within 14 days of randomization)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or calculated creatinine clearance (CrCl) >= 40 mL/min (Cockcroft and Gault or Wright formula may be used according to local practice) (obtained within 14 days of randomization)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x institutional ULN
* Total Bilirubin =< 1.5 x institutional ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for four months after the last dose of pembrolizumab.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG])
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men who are sexually active with WOCBP will be instructed to adhere to contraception for a period of four months after the last dose of investigational product

Exclusion Criteria:

* Requirement of immunosuppressive therapy within 14 days of randomization
* Salivary gland carcinomas, lip carcinoma, adenocarcinoma of the skin
* Prior use of immune checkpoint blockade agent
* History of human immunodeficiency virus (HIV), hepatitis B, C: Participants who test positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection, those who test positive for human immunodeficiency virus (HIV) or have known acquired immunodeficiency syndrome (AIDS)
* Unresectable disease, as determined by the surgeon and team
* Subjects with history of grade 3 toxicity with prior immunotherapy
* Patients with distant metastases
* Subjects with active autoimmune disease
* Breastfeeding women
* Additional prior malignancy within the previous 3 years (treated or untreated, except for skin carcinomas treated with excision alone and carcinoma in situ of the cervix)
* Palliative radiotherapy less than 14 days prior to first dose of study drug
* Any history of hypersensitivity to any of the trial medications
* Poorly controlled or serious medical or psychiatric illness likely to interfere with participation and/or compliance in this clinical trial
* Prisoners or subjects who are involuntarily incarcerated
* Patients not available for follow-up/future contact as defined in the ICF
* Note: Patients on this protocol are not excluded from participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 100 days after last dose of study drug
  Evaluated using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0. Summarized by treatment group. All on-study adverse events (AEs), treatment-related AEs, serious (S)AEs, and treatment-related SAEs will be tabulated using worst grade per NCI CTCAE version 4.0 criteria by system organ class and preferred term. On-study lab parameters including hematology, chemistry, liver function, and renal function will also be summarized using worst grade NCI CTCAE v 4.0 criteria. Toxicity will be measured as the rate of grade 3 and 4 adverse events and will be calculated through using the exact binomial distribution method with a 2- sided 95% confidence interval.
Health related quality of life | Up to 5 years
  Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30. Analysis will be performed in all randomized participants who have an assessment at baseline and at least one follow-up assessment using linear mixed model for repeated measures to model the changes overtime for each arm.

SECONDARY OUTCOMES:
Objective-response rate (ORR) | Up to 5 years
  ORR including complete response rate, partial response rate, and stable disease rate will be calculated using the exact binomial distribution method with a 2- sided 95% confidence interval among patients who obtain a least one dose of study drug.
Local control rate | From the first day of therapy to the occurrence of a local and/or regional recurrence (whichever comes first), and death from any cause other than distant metastasis, assessed up to 24 months
  Analyses will be conducted using Kaplan-Meier method for each arm. The hazard ratio and corresponding two-sided 95% CI will be estimated using a Cox proportional hazards model, with treatment group as a single covariate.
Overall survival | Up to 5 years
  Analyses will be conducted using Kaplan-Meier method for each arm. The hazard ratio and corresponding two-sided 95% CI will be estimated using a Cox proportional hazards model, with treatment group as a single covariate.
Progression-free survival (PFS) | From the first day of the therapy to the appearance of local or regional recurrence, distant metastases, secondary primary cancer or death from any cause, assessed up to 24 months
  Analyses will be conducted using Kaplan-Meier method for each arm. The PFS medians with 95% confidence intervals (CIs), and PFS at 6, 12, and 24 months with 95% CIs will be estimated a two-sided log-rank test. The hazard ratio and corresponding two-sided 95% CI will be estimated using a Cox proportional hazards model, with treatment group as a single covariate, stratified by the above factors.
PD-L1 expression | Up to 5 years
  A Cox proportional hazards model will be used to test the interaction between PD-L1 expression (positive vs negative) and treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Dukagjin M Blakaj, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu